CLINICAL TRIAL: NCT03086837
Title: The Smart City Active Mobile Phone Intervention (SCAMPI) Study: a Randomized Controlled Trial to Promote Physical Activity Through Active Transportation
Brief Title: The Smart City Active Mobile Phone Intervention (SCAMPI)
Acronym: SCAMPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marie Löf, docent, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-00138
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone based intervention (Experimental): Participants in the intervention group will receive a 12 week mobile phone based program via a mobile phone application specifically designed for this study. The program will include information, advice and strategies to increase active transportation. Feedback will be provided on personal goals.
  Interventions: Behavioral: Mobile phone based intervention
- Control (No Intervention): No information

INTERVENTIONS:
Behavioral: Mobile phone based intervention — Participants will receive supporting messages through a mobile phone based intervention.
  Arms: Mobile phone based intervention

SUMMARY:
Physical inactivity is still a major public health problem. Active transportation i.e. walking or cycling for transport can contribute to greater total physical activity. The specific aim of this study is to evaluate if a 12-week mobile phone application can increase time spent in active transportation (cycling or walking) and in moderate-to-vigorous physical activity in Swedish adults aged 20-65 years.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years of age
* living in Stockholm or its suburbs
* being able to understand Swedish sufficiently well in order to understand the purpose of the study and the content of the intervention

Exclusion Criteria:

* having a disease prohibiting them from participation in moderate physical activity such as walking or cycling

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Total activity and moderate-to-vigorous physical activity | At the end of the intervention which is 12 weeks after baseline
  Accelerometer outputs including time spent in moderate-to-vigorous physical activity

SECONDARY OUTCOMES:
Walkability | At the end of the intervention which is 12 weeks after baseline
  Perception of neighborhood
Active transportation | At the end of intervention which is 12 weeks after baseline
  Time spent walking and cycling in minutes per day
Total activity and moderate-to-vigorous physical activity | At the six month follow-up
  Accelerometer outputs including time spent in moderate-to-vigorous physical activity
Walkability | At the six month follow-up
  Perception of neighborhood
Active transportation | At the six month follow-up
  Time spent walking and cycling in minutes per day

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindqvist AK, Rutberg S, Soderstrom E, Ek A, Alexandrou C, Maddison R, Lof M. User Perception of a Smartphone App to Promote Physical Activity Through Active Transportation: Inductive Qualitative Content Analysis Within the Smart City Active Mobile Phone Intervention (SCAMPI) Study. JMIR Mhealth Uhealth. 2020 Aug 5;8(8):e19380. doi: 10.2196/19380. PMID 32755889
- [Derived] Ek A, Alexandrou C, Soderstrom E, Bergman P, Delisle Nystrom C, Direito A, Eriksson U, Henriksson P, Maddison R, Trolle Lagerros Y, Bendtsen M, Lof M. Effectiveness of a 3-Month Mobile Phone-Based Behavior Change Program on Active Transportation and Physical Activity in Adults: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jun 8;8(6):e18531. doi: 10.2196/18531. PMID 32510462
- [Derived] Ek A, Alexandrou C, Delisle Nystrom C, Direito A, Eriksson U, Hammar U, Henriksson P, Maddison R, Trolle Lagerros Y, Lof M. The Smart City Active Mobile Phone Intervention (SCAMPI) study to promote physical activity through active transportation in healthy adults: a study protocol for a randomised controlled trial. BMC Public Health. 2018 Jul 16;18(1):880. doi: 10.1186/s12889-018-5658-4. PMID 30012116